CLINICAL TRIAL: NCT02347696
Title: Effect of Two Programs of Physical Activity of Different Intensity, Mediterranean Diet and the Combination of Both on NAFLD and Erytrocyte Membrane Lipid Profile.
Brief Title: Diet and Physical Activity on NAFLD and Erytrocyte Membrane Lipid Profile.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, Alberto R Osella, MD, PhD, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NUTRIATT
Record Dates: First submitted 2015-01-21; First posted 2015-01-27 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: NAFLD
Keywords: Diet; Physical Activity; Trial; Lipidomics; Occidental Diseases
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Control (Other): The subjects will follow a diet based on INRAN guidelines without doing any physical activity.
  Interventions: Behavioral: Control
- LGIMD (Other): The subjects will follow a Low Glycemic Index Mediterranean Diet without doing any physical activity.
  Interventions: Behavioral: LGIMD
- Endurance Activity (EA) (Other): The subjects will follow a program of endurance (aerobic) activity (EA) without following a specific diet.
  Interventions: Behavioral: Endurance Activity (EA)
- EA+Resistance Training (RT) (Other): The subjects will follow a program of endurance activity (EA) and resistance training (RT) without following a specific diet.
  Interventions: Behavioral: EA+Resistance Training (RT)
- LGIMD+EA (Other): The subjects will follow a Low Glycemic Index Mediterranean Diet (LGIMD) togheter with a program of endurance activity (EA).
  Interventions: Behavioral: LGIMD+EA
- LGIMD+EA/RT (Other): The subjects will follow a Low Glycemic Index Mediterranean Diet (LGIMD) togheter with a program of endurance activity (EA) and resistance training (RT).
  Interventions: Behavioral: LGIMD+EA/RT

INTERVENTIONS:
Behavioral: Control — Subjects will follow a diet based on INRAN guidelines without doing any physical activity.
  Arms: Control
Behavioral: LGIMD — Subjects will follow a Low Glycemic Index Mediterranean Diet (LGIMD) without doing any physical activity.
  Arms: LGIMD
Behavioral: Endurance Activity (EA) — Subject will follow a program of endurance activity as follows:
  Frequency: 3 times/week Duration: 60 minutes
  Intensity:
  * weeks 1-4: 14.2 kcal*kg-1*week-1;
  * weeks 5-8: 18.9 kcal*kg-1*week-1;
  * weeks 9-12: 23.6 kcal*kg-1*week-1.
  Arms: Endurance Activity (EA)
Behavioral: EA+Resistance Training (RT) — Subject will follow a program of endurance activity as follows:
  Frequency: 3 times/week Duration: 60 minutes
  Intensity (for Endurance activity):
  * weeks 1-4: 14.2 kcal*kg-1*week-1;
  * weeks 5-8: 18.9 kcal*kg-1*week-1;
  * weeks 9-12: 23.6 kcal*kg-1*week-1.
  Resistance activity:
  Muscolation: Training of the bigger muscle groups (chest, shoulders, arms, abdomen, back, glutes and legs);
  * Progression: increase of 1-2.5 kg*week-1
  * Training of all muscle groups in the same session
  Arms: EA+Resistance Training (RT)
Behavioral: LGIMD+EA — Subjects will follow a Low Glycemic Index Mediterranean Diet together with a program of endurance activity.
  Arms: LGIMD+EA
Behavioral: LGIMD+EA/RT — Subjects will follow a Low Glycemic Index Mediterranean Diet together with a program of both endurance activity and resistance training.
  Arms: LGIMD+EA/RT

SUMMARY:
This study aims to evaluate the effect of two programs of different intensity level of physical activity, of low glycemic index Mediterranean Diet and of the interaction of both, on NAFLD score and on the lipid composition of the erythrocyte membrane.

DETAILED DESCRIPTION:
The surveys conducted on the populations of Castellana Grotte and Putignano (Bari, Italy) evidenced that Non-Alcoholic Fatty liver Disease (NAFLD) reaches a prevalence of 30%, especially among aged and male individuals. Being a crucial outcome of several metabolic alterations, it becomes imperative for Public Health to adopt strategies aimed to control the factors responsible for NAFLD onset.

The objective of this study is to evaluate the effect of two programs of different intensity level of physical activity, of low glycemic index Mediterranean Diet and of the interaction of both, on NAFLD score and on the lipid composition of the erythrocyte membrane.

Study participants responding to the inclusion criteria of this trial will be chosen both in the hospital setting and in the general practitioners' clinics. At the enrollement, anthropometric and biochemical variables will be measured, as well as bioimpedenziometric and calorimetric parameters; participants will also undergo Fibroscan-CAP to measure the outcome and will be asked about their medical history and life-style. Subjects will be randomized to the different arms of the trial and be followed-up at the end of the sixth and the twelfth week of enrollement.

All data will be statistically analysed by applying the Chi-Square test and t-test for discrete and continuous variables, respectively. As it deals with the analysis of data repeatedly measured on the same subject, the Generalized Estimating Equation (GEE) will be applied to evaluate the effect of the intervention on the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 25.0
* Moderate or severe NAFLD
* 30 < age <60

Exclusion Criteria:

* Overt cardiovascular disease and revascularization procedures;
* Stroke;
* Clinical peripheral artery disease;
* Type-2 Diabetes Mellitus (current treatment with insulin or oral hypoglycemic drugs, fasting glucose >126 mg/dl, or casual glucose >200 mg/dl);
* Severe medical condition that may impair the person to participate in a nutritional intervention study;
* Impossibility to follow Mediterranean Diet for religious or other reasons.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Non-Alcoholic Fatty liver Disease (NAFLD) score | up to 12 weeks
  NAFLD score will be built with Fobroscan-CAP

SECONDARY OUTCOMES:
Lipid composition of erythrocyte membrane | 6 and 12 weeks
Sierical lipid profile | 6 and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alberto R Osella, MD, PhD, Principal Investigator — IRCCS "Saverio De Bellis"
Locations (1):
- Laboratory of Epidemiology and Biostatistics-IRCCS Saverio de Bellis, Castellana Grotte, BA, Italy

IPD SHARING:
Plan to Share IPD: Yes
When data analysis will finish